CLINICAL TRIAL: NCT06729385
Title: The Blood Proteome Profiling Identifies Biomarkers Associated with Prognosis in Ischemic Stroke Due to Large Artery Atherosclerosis
Brief Title: Blood Proteome Profiling Identifies Biomarkers in Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, MD.PhD, Capital Medical University
Other Study IDs: PBIS
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2024-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Obvious group: Patients with large artery atherosclerotic ischemic stroke, presenting 7 to 30 days after onset, and who have not received reperfusion therapy.
  Interventions: Diagnostic Test: The blood Proteome Profiling

INTERVENTIONS:
Diagnostic Test: The blood Proteome Profiling — Patients who meet the inclusion criteria will undergo fasting blood collection for proteomics analysis upon admission.

SUMMARY:
Endovascular thrombectomy and intravenous thrombolysis have become key therapeutic approaches for acute ischemic stroke. However, due to time window limitations, many patients are unable to receive reperfusion therapy, and the majority only receive supportive treatment. Ischemic stroke-related complications, including edema and infection, gradually subside after 7 days post-stroke, with the patient's condition generally stabilizing. Endogenous repair mechanisms will play a critical role in the coming months. This study aims to predict prognostic biomarkers for ischemic stroke patients who have not undergone reperfusion therapy, using blood proteomics data. All samples in our study are derived from this experiment. Our goal is to elucidate the molecular mechanisms underlying post-reperfusion prognosis and to provide insights for optimizing stroke treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18.
* Clinical signs consistent with acute ischemic stroke (TOAST classification: large artery atherosclerosis)
* 7 to 30 days from symptom onset.

Exclusion Criteria:

* Severe infection or multiple organ failure.
* Untreated moderate or severe coronary artery stenosis, or a history of coronary artery bypass surgery.
* Ongoing hemodialysis or peritoneal dialysis, or severe renal insufficiency characterized by a glomerular filtration rate (GFR) of less than 30 ml/min or serum creatinine levels exceeding 220 mmol/L (2.5 mg/dl).
* Known intracranial aneurysm or cerebral arteriovenous malformation.
* Malignant brain tumor or central nervous system (CNS) infection.
* Pre-existing neurological or psychiatric conditions that could confound the neurological or functional assessments.
* Baseline platelet count <50 × 109/L.
* Pregnancy or lactation at the time of admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with large artery atherosclerotic ischemic stroke, presenting 7 to 30 days after onset, and who have not received reperfusion therapy.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measures: | 3 months
  Modified Rankin Scale score (mRS) at 90 days The Modified Rankin Scale (mRS) at 90 days was used to assess functional outcomes. The mRS is a widely utilized scale to measure the degree of disability or dependence in daily activities among stroke patients.
  Minimum value: 0 (indicating no symptoms or disability) Maximum value: 6 (indicating death) Interpretation: Higher scores represent worse outcomes, reflecting greater levels of disability or mortality.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Xuanwu Hospital, Beijing, Beijing Municipality
  - People's hospital of Xiushan Country, Chongqing, Chongqing Municipality
  - Nanyang Nanshi Hospital, Nanyang, Henan
  - Liuyang Jili Hospital, Hunan, China, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No